CLINICAL TRIAL: NCT02011958
Title: A Randomized Trial of Ambisome Monotherapy and Combination of Ambisome and Miltefosine for the Treatment of VL in HIV Positive Patients in Ethiopia Followed by Secondary VL Prophylactic Treatment With Pentamidine.
Brief Title: Efficacy Trial of Ambisome Given Alone and Ambisome Given in Combination With Miltefosine for the Treatment of VL HIV Positive Ethiopian Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Medecins Sans Frontieres, Netherlands (Other); London School of Hygiene and Tropical Medicine (Other); Addis Ababa University (Other); Institute of Tropical Medicine, Belgium (Other); Slotervaart Hospital (Other); University of Gondar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIV/VL 0511
Record Dates: First submitted 2013-11-18; First posted 2013-12-16 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Visceral Leishmaniasis
Keywords: Visceral Leishmaniasis; HIV positive patients; Phase III trial; Randomised; Liposomal amphotericin B; Ambisome; Miltefosine; Pentamidine; Efficacy; Safety
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — liposomal amphotericin B; miltefosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liposomal Amphotericin B / Miltefosine (Experimental): Liposomal Amphotericin B : 30mg/kg total dose: IV infusion 5mg/kg per day on day 1, 3, 5, 7, 9, 11
  Miltefosine: orally taken every day during 28 days
  * 1 x 50 mg capsule per day if patient weights less or equal to 25 kg
  * 2 x 50 mg capsules per day if the patient weights more than 25 kg
  Interventions: Drug: Liposomal Amphotericin B; Drug: Miltefosine
- Liposomal Amphotericin B (Experimental): Liposomal Amphotericin B: 40 mg/kg total dose : IV infusion of 5mg/kg per day on day 1 to 5, 10, 17, 24
  Interventions: Drug: Liposomal Amphotericin B

INTERVENTIONS:
Drug: Liposomal Amphotericin B — 40 mg/kg total dose: IV infusion of 5mg/kg per day on day 1 to 5, 10,17,24 (when administered as a monotherapy)
  30 mg/kg total dose: IV infusion 5 mg/kg per day on day 1, 3, 5, 7, 9, 11 (when administered in combination with Miltefosine)
  Other Names: Ambisome
Drug: Miltefosine — Orally taken every day during 28 days
  * 1 x 50 mg capsule per day if the patient weights less or equal to 25 kg
  * 2 x 50 mg capsules per day if the patient weights more than 25 kg (1 capsule in the morning / 1 capsule in the evening)
  Other Names: Impavido
  Arms: Liposomal Amphotericin B / Miltefosine

SUMMARY:
The overall objective of this trial is to identify a safe and effective treatment for visceral leishmaniasis (VL) in HIV co-infected Ethiopian patients.

Patients will receive either Ambisome alone or Ambisome in combination with Miltefosine.

Patients who do not undergo treatment failure will be given a VL prophylactic treatment with Pentamidine one month after the end of the study treatment.

DETAILED DESCRIPTION:
Visceral Leishmaniasis (VL) is a neglected disease which is fatal if left untreated. Ethiopia is one of the countries where the majority of cases occur. With spread of HIV in VL endemic areas an increase in co-infected cases has been reported in Ethiopia.

HIV and VL mutually influence each other as they both affect cellular immunity. The most important features of co-infection include poor outcome, increased drug toxicity and relapse of treatment with the need for maintenance therapy.

There are few studies in co-infected patients. There are no specific recommendations for HIV-VL co-infected patients in Ethiopia.

This protocol will evaluate the efficacy and safety of the combination of Ambisome with Miltefosine and Ambisome monotherapy (high dose) in Ethiopia.

It is designed as a randomised, parallel arm, open-label trial. No comparator will be included.

The randomization will be stratified according to centre as well as wether VL is a primary case or a relapse. The study will be analysed according to group-sequential methods, specifically the triangular test. Data from each arm will be analysed after every 10 patients reach the primary endpoint of final cure at day 29. The data will be analysed as proportions according to an intention to treat and per protocol analysis for each arm.In order to address potential heterogeneity of the population, a test will be performed when a treatment is stopped. Depending on the outcome of this test for heterogeneity, recruitment may be continued into one stratum.

The treatment duration will be 28 days or 56 days in case of extended treatment.

* If at Day 29 assessment, tissue aspirate is parasite negative, the patient will be eligible for secondary prophylaxis (Pentamidine 4mg/kg IM (intramuscular) once a month up to a maximum of 18 months) and enter the 1 year follow up phase.
* If at day 29 assessment, tissue aspirate is positive but the patient is well, he/she will receive another complete course of treatment (but classified as treatment failure). The patient will be evaluated again on day 58. Those who still have a parasite positive tissue aspirate will be offered a rescue treatment. Those who are negative will be offered secondary prophylaxis if eligible (Pentamidine 4mg/kg IM once a month up to a maximum of 18 months).
* If at day 29 assessment, tissue aspirate is positive and the patient is unwell, he/she will be treated with rescue treatment (and considered as treatment failure)
* All patients, independently of their outcome at day 29 and/or day 58 will enter the follow-up assessments at day 210 and day 390.

Rescue treatment will also be given in case of relapse during the follow-up period and in case of occurence of severe grade 2 or grade 3 PKDL or PKDL with mucosal and/or eye involvement after treatment period.

All patients who are not yet on antiretroviral treatment (ART) at inclusion will commence ART once they have completed routine voluntary counselling and testing procedures. Patients who are already on ART at diagnosis of VL will continue ART throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV positive test (2 rapid diagnostics tests (RDTs) followed by a confirmatory ELISA test).
* Diagnosis of VL (first episode or relapse) confirmed by bone marrow or spleen aspirate.
* Male and female age: 18-60 years.
* Written informed consent from the patient.

Exclusion Criteria:

* Women of child-bearing potential (defined as women who have achieved menarche) who are not using an assured method of contraception or are unwilling to use an assured method of contraception for the duration of treatment and four months after.
* Pregnant women or breast-feeding mothers.
* Patients with grade 2 or 3 post kala-azar dermal leishmaniasis (PKDL) lesions.
* Clinical or biological evidence of severe cardiac, renal or hepatic impairment.
* Known hypersensitivity to AmBisome® and/or miltefosine.
* Patients receiving allopurinol treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Initial parasitological cure at day 29 | Day 29
  Absence of parasites in tissue aspirate at day 29; hence no rescue medication provided up to this time-point.

SECONDARY OUTCOMES:
Relapse-free survival at day 390 | Day 390
  The patient being alive and disease free from day 29 (if initially cured) or day 58 in case of extended treatment (absence of signs and symptoms of visceral leishmaniasis or if symptomatic, a negative parasitological assessment by tissue aspirate)

OTHER OUTCOMES:
Safety endpoint | From the first dose of study medication up to 1 month after the stop of treatment
  Adverse Events and Serious Adverse Events
Response to antiretroviral treatment | Screening , Day 29, Day 58, Day 210 and Day 390
  Measurement of CD4 (cluster of differentiation 4) count and HIV viral load
Pharmacokinetics: drug-drug interaction between VL treatment and antiretroviral drugs (Arm 1: PK AmphoB (Amphotericin B) and PK/EFV (Efavirenz)/NVP (Nevirapine)/LPV (Lopinavir)/RTV, Arm 2: PK AmphoB, PK Miltefosine and PK EFV/NVP/LPV/RTV) | Arm1:PK AmphoB, Day 1 and 24 post-dose / PK EFV/NVP/LPV/RTV: Day 1,24,58,210 and 390 post-dose. Arm 2: PK AmphoB, Day 1 and 11 post-dose/PK Miltefosine: Pre-dose, day 11,29,58,210 post-dose / PK EFV/NVP/LPV/RTV: Day 1,29,58,210 and 390 post-dose
  In a subgroup of patients, blood concentrations of Ambisome (EDTA plasma), Miltefosine (DBS) and Anti Retroviral Drugs (DBS)

CONTACTS AND LOCATIONS:
Overall Officials: Ermias Diro, Dr. MD, Principal Investigator — University of Gondar
Locations (2):
- Ethiopia (2):
  - MSF, Abdurafi
  - Leishmaniasis Research Center, University Hospital of Gondar, Gonder

REFERENCES:
- [Result] Diro E, Blesson S, Edwards T, Ritmeijer K, Fikre H, Admassu H, Kibret A, Ellis SJ, Bardonneau C, Zijlstra EE, Soipei P, Mutinda B, Omollo R, Kimutai R, Omwalo G, Wasunna M, Tadesse F, Alves F, Strub-Wourgaft N, Hailu A, Alexander N, Alvar J. A randomized trial of AmBisome monotherapy and AmBisome and miltefosine combination to treat visceral leishmaniasis in HIV co-infected patients in Ethiopia. PLoS Negl Trop Dis. 2019 Jan 17;13(1):e0006988. doi: 10.1371/journal.pntd.0006988. eCollection 2019 Jan. PMID 30653490
- [Result] Diro E, Edwards T, Ritmeijer K, Fikre H, Abongomera C, Kibret A, Bardonneau C, Soipei P, Mutinda B, Omollo R, van Griensven J, Zijlstra EE, Wasunna M, Alves F, Alvar J, Hailu A, Alexander N, Blesson S. Long term outcomes and prognostics of visceral leishmaniasis in HIV infected patients with use of pentamidine as secondary prophylaxis based on CD4 level: a prospective cohort study in Ethiopia. PLoS Negl Trop Dis. 2019 Feb 21;13(2):e0007132. doi: 10.1371/journal.pntd.0007132. eCollection 2019 Feb. PMID 30789910